CLINICAL TRIAL: NCT06447519
Title: Clinical and Radiographic Outcomes of Multiple-Visit Non-Surgical Root Canal Treatment in Permanent Teeth With Symptomatic Apical Periodontitis : Interappointment Dressing or Not? A Randomized Clinical Trial
Brief Title: Multiple-Visit RCT in Teeth With SAP: Interappointment Dressing or Not?
Acronym: RCTCa(OH)2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 230/21-03-2024
Record Dates: First submitted 2024-05-27; First posted 2024-06-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Endodontically Treated Teeth; Calcium Hydroxide
Keywords: Multivisit Endodontic Treatment; Interapointment dressing; Apical Periodontitis; Outcome
MeSH Terms: conditions — Tooth, Nonvital; Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ca(OH)2 intracanal medicament (Experimental): Ca(OH)2 intracanal medicament used for root canal disinfection as interapointment dressing.
  Interventions: Drug: Ca(OH)2 as intracanal medicament
- Standard of Care (No Intervention): No intracanal medicament. The root canal will be left empty without any intracanal dressing between appointments.

INTERVENTIONS:
Drug: Ca(OH)2 as intracanal medicament — Ca(OH2 will be used as intracanal medicament for the disinfection of the root canal between appointmnents
  Arms: Ca(OH)2 intracanal medicament

SUMMARY:
The aim of the study is to evaluate the effectiveness of calcium hydroxide as an intracanal medicament in the clinical and radiographic healing of periapical tissues in teeth diagnosed with symptomatic apical periodontitis. This evaluation will be conducted after multiple visit endodontic treatment. The follow-up sessions will be programmed from 6 to 24 months postoperatively. Postoperative pain will also be considered as a secondary outcome. Participants will be asked to rate their pain level on a numerical scale from 0 to10 before and after each session of endodontic treatment. Additionally, the use of analgesics after the procedure will be measured and the incidence of flare-ups will be evaluated. Two study groups will be formed to undergo multiple-visit endodontic treatment. The intervention group will receive intracanal medication of calcium hydroxide, while the control group will have the root canal left empty between appointments.

DETAILED DESCRIPTION:
The first visit will include the following clinical steps . After administering local anesthesia with 4% articaine hydrochloride and epinephrine injection (with 1:200,000 adrenaline) or 2% mepivacaine for an inferior alveolar block, all decayed tissue from the tooth will be removed. The tooth will be isolated with a rubber dam, the tooth crown will be disinfected with 2% NaOCl, and an access cavity preparation will be created. The #10 C-Pilot file will be used to create a glide path. The working length will be established with an apex locator and an x-ray. The root canal will be instrumented using the sequence of NiTi rotary files Edge Endo X7. The canals will be irrigated copiously with 10ml of 2% NaOCl each time. Following instrumentation, a final rinse with 10ml of 2% NaOCl, 10ml of 17% EDTA, and 10ml of saline solution will be performed. Group 1 will receive intracanal dressing with Ca (OH)2 paste using Lentulo for a period of 7-10 days. Group 2 will be left without intracanal dressing for a period of 7-10 days. In both groups, teeth will be restored with glass ionomer cement (GIC) as a temporary restoration. The final visit will include the following clinical steps. After examining the tooth and surrounding tissues, local anesthesia will be administered as previously described. The temporary restorative material will be removed, and the tooth will be isolated with a rubber dam before accessing the root canal. In Group 1, the intracanal dressing will be removed through irrigation, and then obturated using a standardized, matched size and taper gutta-percha cone with AH-plus sealer with the single-cone obturation technique. The tooth will be then temporarily restored with glass ionomer cement (GIC), and the participant will be referred for final restoration within 7-14 days. The same protocol is followed for Group 2.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade: I or II
* Age: ≥18 years
* Permanent teeth
* Pulp diagnosis: necrosis or previously treated
* Diagnosis of periapical tissues: symptomatic apical periodontitis
* Teeth sensitive to percussion and/or palpation
* Initial PAI: 3-5
* Signed Patient Consent Statement for participation in clinical research

Exclusion Criteria:

* Subjects that do not meet the inclusion criteria
* Pregnant women
* Patients who receive corticosteroids and/or have received antibiotics within the previous three months
* Patients who report pain in a different area than that of the tooth under investigation
* Teeth that cannot be isolated with a rubber dam
* Teeth with extensive hard tissue destruction that is not restorable
* Teeth with an anatomic peculiarity of the root canal (internal resorption, perforation, displacement of root canal course due to previous endodontic treatment)
* Teeth in which the formation of the apex has not been completed
* Fractured teeth with periodontal involvement
* Teeth with periodontal pocket depth ≥ 4mm or teeth with bone loss at the bifurcation of the roots due to periodontitis
* Teeth with loss of periodontal attachment ≥ 5 mm
* Teeth with embedded exudate in the session planned for root canal obturation.
* Teeth that after completion of the endodontic treatment show underocclusion >2mm or hyperobstruction >1mm from the radiographic apex.
* Teeth in which permanent restoration has not been completed over time less than one month after endodontic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09-12 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
Clinical evidence of success | 6-24 months post-operatively
  Criteria of clinical success include the absence of pain and tenderness to palpation and percussion and the absence of sinus or any associated soft tissue swelling. Failure is indicated by the presence of at least one of the abovementioned signs or symptoms.
Radiographic evidence of success | 6-24 months post-operatively
  Radiographic evidence of periapical healing will be evaluated by the improvement of Periapical Index score (PAI). The PAI system provides an ordinal scale of 5 scores ranging from 1 (healthy) to 5 ( severe periodontitis with exacerbating features). In detail PAI score 1 indicates normal periapical anatomy. PAI score 2 indicates mild changes in bone pattern. PAI score 3 is indicative by changes in bone pattern with diffuse loss of mineral. PAI score 4 is indicative of apical periodontitis with definite radiolucency in the periapical area. PAI score 5 indicates severe periodontitis with exacerbating features. Improvement of PAI score will be evaluated as success. Consequently a lower PAI score is indicative of success but a higher or stable PAI score is indicative of failure.

SECONDARY OUTCOMES:
Flare-up incidence | 0 to 3 days after every single appointment
  Patients will contact the primary investigator in case of pain or swelling that may appear after each appointment.
Postoperative pain assesment | 0 to 3 days after every single appointment
  Description: Participants will be advised to follow analgesic medication of Ibuprofen (600mg) or Paracetamol (1000mg) treatment or combined medication only in case of feeling pain. Participants will be asked to rate the level of pain on a numerical rating scale from 0 to10 before the start and after 1, 2 and 3 days of each session. According to this scale 0 is indicative of "no pain" and 10 is indicative of "the worst pain ever felt". All intermediate scales are proportional to the pain of the patient. For example, 1 to 3 is indicative of mild pain, 4 to 6 moderate pain and 7 to 9 severe pain. Participants will also be given a paper form in which they must fill in the type and quantity of receiving analgesic medication for each of the first 3 days after each session of endodontic therapy. Besides the numerical pain scale the number of analgesic tablets will be also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Economides, Prof., Study Director — School of Dentistry, Aristotle University of Thessaloniki
Locations (1):
- School of Dentitry, Aristotle University of Thessaloniki, Thessaloniki, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiger R, Rosendahl R, Lost C. Influence of calcium hydroxide intracanal dressings on the prognosis of teeth with endodontically induced periapical lesions. Int Endod J. 2000 May;33(3):219-26. doi: 10.1046/j.1365-2591.1999.00298.x. PMID 11307438
- [Background] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729
- [Background] Mergoni G, Ganim M, Lodi G, Figini L, Gagliani M, Manfredi M. Single versus multiple visits for endodontic treatment of permanent teeth. Cochrane Database Syst Rev. 2022 Dec 13;12(12):CD005296. doi: 10.1002/14651858.CD005296.pub4. PMID 36512807
- [Background] Rossi-Fedele G, Rodig T. Effectiveness of root canal irrigation and dressing for the treatment of apical periodontitis: A systematic review and meta-analysis of clinical trials. Int Endod J. 2023 Oct;56 Suppl 3:422-435. doi: 10.1111/iej.13777. Epub 2022 May 31. PMID 35579074
- Available data/document: Study Protocol — https://ikee.lib.auth.gr — https://ikee.lib.auth.gr